CLINICAL TRIAL: NCT03963999
Title: Validating Ultrasound Biomarkers for Hepatic Sinusoidal Obstruction Syndrome in Pediatric Hematopoietic Cell Transplant Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We did not receive grant funding. We will reapply in June of 2020
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Nationwide Children's Hospital (Other); St. Jude Children's Research Hospital (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000792
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sinusoidal Obstruction Syndrome; Veno Occlusive Disease, Hepatic; Bone Marrow Transplant Complications; Stem Cell Transplant Complications
Keywords: Ultrasound Elastography
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Intervention Model Description: All patients undergoing myeloblative conditioning regimen as part of hematopoietic cell transplant or prior liver damage or other high risk factor will be consecutively studied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Undergoing HCT (Experimental): All patients enrolled will undergo grayscale US, Doppler US, US SWE and CEUS at specific time points as outlined in the protocol based on disease course.
  Interventions: Diagnostic Test: Ultrasound Elastography; Drug: Contrast Enhanced Ultrasound (CEUS)

INTERVENTIONS:
Diagnostic Test: Ultrasound Elastography — Ultrasound shear wave elastography
Drug: Contrast Enhanced Ultrasound (CEUS) — Contrast-enhanced ultrasound (CEUS) uses an intravenous injection of microbubble contrast agent.
  Other Names: Lumason (sulfur hexafluoride lipid-type A microspheres)

SUMMARY:
Hepatic veno-occlusive disease/sinusoidal obstructive syndrome (VOD/SOS) is a potentially fatal complication of hematopoietic cell transplant (HCT). Historically VOD/SOS has been clinically diagnosed using the modified Seattle criteria or the Baltimore criteria. The modified Seattle Criteria define VOD/SOS diagnosis is made when two of the following three criteria are present in a patient within 21 days of transplantation: hyperbilirubinemia (total serum bilirubin > 2 mg/dL), hepatomegaly or right upper quadrant liver pain, and weight gain (> 2% of baseline) or ascites. Other conditions like graft versus host disease, sepsis syndrome (fever and hypotension), cardiac failure, or tumor infiltration) have to be excluded. This definition was from a well-designed retrospective cohort study on 255 adult and pediatric HCT patients in which the VOD/SOS incidence was 21%. McDonald et al followed up this work with a prospective cohort study of 355 patients noting an incidence of VOD/SOS of 54%. These seminal studies have had a major impact on the field by defining clinical diagnostic criteria. An alternative diagnostic criteria (Baltimore criteria) was proposed by Jones et al as a part of a well-designed retrospective review of 235 HCT patients finding a VOD/SOS incidence of 22%. Jones defined VOD/SOS as the presence of hyperbilirubinemia (total serum bilirubin > 2 mg/dL) along with at least 2 of 3 other findings: hepatomegaly, ascites, and weight gain (> 5% of baseline).

DETAILED DESCRIPTION:
Hepatic veno-occlusive disease/sinusoidal obstructive syndrome (VOD/SOS) is a potentially fatal complication of hematopoietic cell transplant (HCT). Historically VOD/SOS has been clinically diagnosed using the modified Seattle criteria or the Baltimore criteria. The modified Seattle Criteria define VOD/SOS diagnosis is made when two of the following three criteria are present in a patient within 21 days of transplantation: hyperbilirubinemia (total serum bilirubin > 2 mg/dL), hepatomegaly or right upper quadrant liver pain, and weight gain (> 2% of baseline) or ascites. Other conditions like graft versus host disease, sepsis syndrome (fever and hypotension), cardiac failure, or tumor infiltration) have to be excluded. This definition was from a well-designed retrospective cohort study on 255 adult and pediatric HCT patients in which the VOD/SOS incidence was 21%. McDonald et al followed up this work with a prospective cohort study of 355 patients noting an incidence of VOD/SOS of 54%. These seminal studies have had a major impact on the field by defining clinical diagnostic criteria. An alternative diagnostic criteria (Baltimore criteria) was proposed by Jones et al (1987) as a part of a well-designed retrospective review of 235 HCT patients finding a VOD/SOS incidence of 22%. Jones defined VOD/SOS as the presence of hyperbilirubinemia (total serum bilirubin > 2 mg/dL) along with at least 2 of 3 other findings: hepatomegaly, ascites, and weight gain (> 5% of baseline).

A large well-executed meta-analysis on 24,920 adults and pediatric patients confirms the fact that applying the more stringent Baltimore criteria results in a lower incidence rate for VOD/SOS of 9.6% as compared to 17.3% with the modified Seattle criteria. A major weakness of this large meta-analysis is that it did not perform a separate pediatric incidence. A small retrospective cohort study of 142 pediatric patients (Barker et al, BMT 2003) reported an incidence of 18% using the modified Seattle criteria corroborating the findings from the meta-analysis.

VOD/SOS is important to study because the survival rates in severe disease with multi-organ failure are very low. Day 100 (post HCT) survival rate for severe VOD/SOS in the meta-analysis was only 16%; most patients died of multi-organ failure. Fortunately, defibrotide seems to be effective in increasing survival rates. Richardson et al (2016) demonstrated in a well-designed and executed phase 3 clinical trial that defibrotide increased day 100 survival in severe VOD/SOS (defined by the Baltimore criteria) with multi-organ failure from 25% to 38%. Weaknesses of this study were that it only included 44 pediatric patients and a historical cohort was used as the control population. A well-designed small, multi-institution, retrospective cohort study in 45 pediatric patients diagnosed with VOD/SOS showed that the complete response rate was 83% in the cohort who started defibrotide treatment within two days of diagnosis and the complete response rate decreased to 10% in patients who started treatment three or more days after clinical diagnosis. A large, well conducted and executed trial of defibrotide involving 101 centers in the USA was also able to confirm this survival benefit. In the 570 pediatric (< 16 years old) patients in this study, the estimated day 100 survival rate was 67.9%. In 512 pediatric and adult patients with VOD/SOS with multi-organ failure, the estimated survival rate was 49.5%. This large study also showed that earlier initiation of defibrotide was associated with increased survival, especially if treatment could be initiated within day 2 after diagnosis. This study lacked a control arm for comparison but historical data showing a survival rate of 16% can again serve as a control here.

In 2017 the European society for Blood and Marrow Transplantation (EBMT) consortium proposed VOD/SOS diagnostic and severity grading criteria specifically for children, which are not distinguished as separate in the Baltimore or Seattle criteria (Corbacioglu et al, 2017). These criteria highlight how VOD/SOS in children differs from adults. Unlike the Baltimore or modified Seattle criteria, EBMT criteria have no time limitation for the diagnosis. The EBMT criteria reinforces the fact that hyperbilirubinemia in children is a late finding. The EBMT proposed grading of severity into four categories: mild, moderate, severe and very severe VOD/SOS. Defibrotide has been investigated and has shown benefit primarily as treatment for VOD/SOS with multi-organ failure, which corresponds to severe and very severe disease by the EBMT severity grading. The weakness of these criteria is that they are not yet tested, but this is something we also aim to do with the proposed research. One of the greatest clinical challenges is determining which patients will progress to severe disease, so that specific therapy can be initiated early. Currently, no clinical, laboratory or imaging biomarkers can reliably differentiate VOD/SOS from other HCT complications. Additionally, there is no biomarker that can reliably differentiate VOD/SOS patients who will go on to develop severe or very severe disease versus VOD/SOS patients who never progress to those severe disease states. Therefore, this research is timely because the investigator's preliminary data reviewed below show that promising imaging biomarkers may be available that can diagnose VOD/SOS earlier than current clinical criteria. These biomarkers could help refine the clinical criteria to allow earlier diagnosis of VOD/SOS, thereby allowing earlier initiation of specific therapy which can help decrease the high mortality from severe VOD/SOS. Additionally, if these biomarkers could identify the VOD/SOS patients at risk of progression to severe or very severe VOD/SOS, this therapy could even be more targeted.

Data Collection Procedures: Candidates for the study will be identified by a HCT physician taking care of the patient and will be identified as a potential candidate for the study. Subjects will be approached for consent by a member of the research team prior to start of conditioning regimen. Consented subjects will have demographic, laboratory and clinical data collected from the chart at each ultrasound time point.

Consented subjects will have grayscale US, Doppler US, US SWE and CEUS within 30 days prior to starting their conditioning regimen.

US Schedule (All exams can be performed +/- 2 days compared to the prescribed date):

Baseline exam: one time within 30 days before start of conditioning (~Day -9).

Inpatient exams: Day -3, day +3, day +7, day + 10, day +17, day +24, day +31, day +60 and day +90 after HCT.

If the patient is discharged earlier than day +100 from the HCT admission, then all exams after the discharge day will be canceled.

Concern for VOD/SOS:

If the HCT team is suspecting VOD/SOS a patient admitted for HCT, then US will be performed twice a week during the time of concern for VOD/SOS.

ELIGIBILITY:
Inclusion Criteria:

* HCT patient under 25 years of age with
* myeloablative conditioning,
* prior liver damage or
* other high risk factor:
* Neuroblastoma,
* HLH,
* Osteopetrosis,
* Thalassemia,
* Treatment with inotuzumab or gemtuzumab within 3 months prior to HCT admission,
* Hepatic iron overload,
* Steatohepatitis,
* Active inflammatory or infection hepatitis or
* Any other condition which puts the patient at a higher risk of developing VOD).

Exclusion Criteria:

* Any patient who has contraindication to any of the ultrasound procedures (e.g. unable to hold still).

Ages: 1 Month to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Define Sensitivity and Specificity of US (grayscale, Doppler and SWE) for Diagnosis and Severity Grading for SOS/VOD | 100 days post transplant
  Determine the sensitivity and specificity of US for diagnosis and severity grading of VOD/SOS in a cohort of 250 pediatric HCT patients.
Define Sensitivity and Specificity of CEUS for Diagnosis and Severity Grading for SOS/VOD | 100 days post transplant
  Determine the sensitivity and specificity of contrast enhanced ultrasound (CEUS) variables for diagnosis and severity grading of VOD/SOS as compared to the pediatric EBMT criteria.
Define Optimal Timing for US for Early Diagnosis and Risk Stratification of VOD/SOS | 100 days post transplant
  Determine the optimal timing for ultrasound measurements to help predict early diagnosis and risk stratification of VOD/SOS.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin S Chan, MD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr RG, Ferraioli G, Palmeri ML, Goodman ZD, Garcia-Tsao G, Rubin J, Garra B, Myers RP, Wilson SR, Rubens D, Levine D. Elastography Assessment of Liver Fibrosis: Society of Radiologists in Ultrasound Consensus Conference Statement. Radiology. 2015 Sep;276(3):845-61. doi: 10.1148/radiol.2015150619. Epub 2015 Jun 16. PMID 26079489
- [Background] Barker CC, Butzner JD, Anderson RA, Brant R, Sauve RS. Incidence, survival and risk factors for the development of veno-occlusive disease in pediatric hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2003 Jul;32(1):79-87. doi: 10.1038/sj.bmt.1704069. PMID 12815482
- [Background] Colecchia A, Ravaioli F, Sessa M, Alemanni VL, Dajti E, Marasco G, Vestito A, Zagari RM, Barbato F, Arpinati M, Cavo M, Festi D, Bonifazi F. Liver Stiffness Measurement Allows Early Diagnosis of Veno-Occlusive Disease/Sinusoidal Obstruction Syndrome in Adult Patients Who Undergo Hematopoietic Stem Cell Transplantation: Results from a Monocentric Prospective Study. Biol Blood Marrow Transplant. 2019 May;25(5):995-1003. doi: 10.1016/j.bbmt.2019.01.019. Epub 2019 Jan 18. PMID 30660772
- [Background] Coppell JA, Richardson PG, Soiffer R, Martin PL, Kernan NA, Chen A, Guinan E, Vogelsang G, Krishnan A, Giralt S, Revta C, Carreau NA, Iacobelli M, Carreras E, Ruutu T, Barbui T, Antin JH, Niederwieser D. Hepatic veno-occlusive disease following stem cell transplantation: incidence, clinical course, and outcome. Biol Blood Marrow Transplant. 2010 Feb;16(2):157-68. doi: 10.1016/j.bbmt.2009.08.024. Epub 2009 Sep 18. PMID 19766729
- [Background] Corbacioglu S, Carreras E, Ansari M, Balduzzi A, Cesaro S, Dalle JH, Dignan F, Gibson B, Guengoer T, Gruhn B, Lankester A, Locatelli F, Pagliuca A, Peters C, Richardson PG, Schulz AS, Sedlacek P, Stein J, Sykora KW, Toporski J, Trigoso E, Vetteranta K, Wachowiak J, Wallhult E, Wynn R, Yaniv I, Yesilipek A, Mohty M, Bader P. Diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in pediatric patients: a new classification from the European society for blood and marrow transplantation. Bone Marrow Transplant. 2018 Feb;53(2):138-145. doi: 10.1038/bmt.2017.161. Epub 2017 Jul 31. PMID 28759025
- [Background] Corbacioglu S, Greil J, Peters C, Wulffraat N, Laws HJ, Dilloo D, Straham B, Gross-Wieltsch U, Sykora KW, Ridolfi-Luthy A, Basu O, Gruhn B, Gungor T, Mihatsch W, Schulz AS. Defibrotide in the treatment of children with veno-occlusive disease (VOD): a retrospective multicentre study demonstrates therapeutic efficacy upon early intervention. Bone Marrow Transplant. 2004 Jan;33(2):189-95. doi: 10.1038/sj.bmt.1704329. PMID 14661036
- [Background] Fontanilla T, Hernando CG, Claros JC, Bautista G, Minaya J, Del Carmen Vega M, Piazza A, Mendez S, Rodriguez C, Aranguena RP. Acoustic radiation force impulse elastography and contrast-enhanced sonography of sinusoidal obstructive syndrome (Veno-occlusive Disease): preliminary results. J Ultrasound Med. 2011 Nov;30(11):1593-8. doi: 10.7863/jum.2011.30.11.1593. PMID 22039033
- [Background] Jones RJ, Lee KS, Beschorner WE, Vogel VG, Grochow LB, Braine HG, Vogelsang GB, Sensenbrenner LL, Santos GW, Saral R. Venoocclusive disease of the liver following bone marrow transplantation. Transplantation. 1987 Dec;44(6):778-83. doi: 10.1097/00007890-198712000-00011. PMID 3321587
- [Background] Kernan NA, Grupp S, Smith AR, Arai S, Triplett B, Antin JH, Lehmann L, Shore T, Ho VT, Bunin N, Iacobelli M, Liang W, Hume R, Tappe W, Soiffer R, Richardson P. Final results from a defibrotide treatment-IND study for patients with hepatic veno-occlusive disease/sinusoidal obstruction syndrome. Br J Haematol. 2018 Jun;181(6):816-827. doi: 10.1111/bjh.15267. Epub 2018 May 16. PMID 29767845
- [Background] Kernan NA, Richardson PG, Smith AR, Triplett BM, Antin JH, Lehmann L, Messinger Y, Liang W, Hume R, Tappe W, Soiffer RJ, Grupp SA. Defibrotide for the treatment of hepatic veno-occlusive disease/sinusoidal obstruction syndrome following nontransplant-associated chemotherapy: Final results from a post hoc analysis of data from an expanded-access program. Pediatr Blood Cancer. 2018 Oct;65(10):e27269. doi: 10.1002/pbc.27269. Epub 2018 Jun 6. PMID 29873895
- [Background] Lassau N, Leclere J, Auperin A, Bourhis JH, Hartmann O, Valteau-Couanet D, Benhamou E, Bosq J, Ibrahim A, Girinski T, Pico JL, Roche A. Hepatic veno-occlusive disease after myeloablative treatment and bone marrow transplantation: value of gray-scale and Doppler US in 100 patients. Radiology. 1997 Aug;204(2):545-52. doi: 10.1148/radiology.204.2.9240551.
- [Background] McDonald GB, Hinds MS, Fisher LD, Schoch HG, Wolford JL, Banaji M, Hardin BJ, Shulman HM, Clift RA. Veno-occlusive disease of the liver and multiorgan failure after bone marrow transplantation: a cohort study of 355 patients. Ann Intern Med. 1993 Feb 15;118(4):255-67. doi: 10.7326/0003-4819-118-4-199302150-00003. PMID 8420443
- [Background] McDonald GB, Sharma P, Matthews DE, Shulman HM, Thomas ED. Venocclusive disease of the liver after bone marrow transplantation: diagnosis, incidence, and predisposing factors. Hepatology. 1984 Jan-Feb;4(1):116-22. doi: 10.1002/hep.1840040121. PMID 6363247
- [Background] Nishida M, Kahata K, Hayase E, Shigematsu A, Sato M, Kudo Y, Omotehara S, Iwai T, Sugita J, Shibuya H, Shimizu C, Teshima T. Novel Ultrasonographic Scoring System of Sinusoidal Obstruction Syndrome after Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2018 Sep;24(9):1896-1900. doi: 10.1016/j.bbmt.2018.05.025. Epub 2018 May 24. PMID 29803752
- [Background] Reddivalla N, Robinson AL, Reid KJ, Radhi MA, Dalal J, Opfer EK, Chan SS. Using liver elastography to diagnose sinusoidal obstruction syndrome in pediatric patients undergoing hematopoetic stem cell transplant. Bone Marrow Transplant. 2020 Mar;55(3):523-530. doi: 10.1038/s41409-017-0064-6. Epub 2018 Jan 15. PMID 29335626
- [Background] Richardson PG, Riches ML, Kernan NA, Brochstein JA, Mineishi S, Termuhlen AM, Arai S, Grupp SA, Guinan EC, Martin PL, Steinbach G, Krishnan A, Nemecek ER, Giralt S, Rodriguez T, Duerst R, Doyle J, Antin JH, Smith A, Lehmann L, Champlin R, Gillio A, Bajwa R, D'Agostino RB Sr, Massaro J, Warren D, Miloslavsky M, Hume RL, Iacobelli M, Nejadnik B, Hannah AL, Soiffer RJ. Phase 3 trial of defibrotide for the treatment of severe veno-occlusive disease and multi-organ failure. Blood. 2016 Mar 31;127(13):1656-65. doi: 10.1182/blood-2015-10-676924. Epub 2016 Jan 29. PMID 26825712
- [Background] Richardson PG, Smith AR, Triplett BM, Kernan NA, Grupp SA, Antin JH, Lehmann L, Miloslavsky M, Hume R, Hannah AL, Nejadnik B, Soiffer RJ. Earlier defibrotide initiation post-diagnosis of veno-occlusive disease/sinusoidal obstruction syndrome improves Day +100 survival following haematopoietic stem cell transplantation. Br J Haematol. 2017 Jul;178(1):112-118. doi: 10.1111/bjh.14727. Epub 2017 Apr 26. PMID 28444784
- [Background] Thumar VD, Vallurupalli VM, Robinson AL, Staggs VS, Shah V, Dalal J, Chan SS. Spectral Doppler Ultrasound Can Help Diagnose Children With Hepatic Sinusoidal Obstructive Syndrome After Hematopoietic Stem Cell Transplantation. Ultrasound Q. 2020 Mar;36(1):6-14. doi: 10.1097/RUQ.0000000000000441. PMID 30921102
- [Background] Trenker C, Wilhelm C, Neesse A, Rexin P, Gorg C. Contrast-Enhanced Ultrasound in Pulmonary Lymphoma: A Small Pilot Study. J Ultrasound Med. 2018 Dec;37(12):2943-2947. doi: 10.1002/jum.14651. Epub 2018 May 6. PMID 29732588